CLINICAL TRIAL: NCT05335876
Title: Long-term Follow-up of Patients With Spinal Muscular Atrophy Treated With OAV101 IT or OAV101 IV in Clinical Trials
Brief Title: Long-term Follow-up of Patients With Spinal Muscular Atrophy Treated With OAV101 in Clinical Trials
Acronym: SPECTRUM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COAV101A12308
Record Dates: First submitted 2022-04-12; First posted 2022-04-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: Zolgensma; OAV101; AVXS 101; gene therapy; Muscle atrophy; SBMA; spinal and bulbar muscular atrophy; spinal muscular atrophy; bulbar muscular atrophy; muscle function; myopathy; muscle wasting; atrophied muscle; loss of muscle strength; Spinal Muscular Atrophy (SMA); survival motor neuron 1 gene (SMN1); SMN protein depletion; survival motor neuron 2 gene (SMN2); chromosome 5q13; neurogenetic disorder; onasemnogene abeparvovec
MeSH Terms: conditions — Muscular Atrophy, Spinal; Muscular Atrophy; Bulbo-Spinal Atrophy, X-Linked; Muscular Diseases | interventions — Zolgensma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous (IV) & Intrathecal (IT) Onasemnogene Abeparvovec (Experimental): Patients who received OAV101 IT or OAV101 IV in clinical trials (COAV101A12306, COAV101B12301 and COAV101B12302)
  Interventions: Biological: onasemnogene abeparvovec

INTERVENTIONS:
Biological: onasemnogene abeparvovec — Onasemnogene abeparvovec is a non-replicating recombinant adeno-associated virus serotype 9 containing the human survival motor neuron gene under the control of the ytomegalovirus enhancer/chicken β-actin-hybrid promoter. Onasemnogene abeparvovec is administered as a one-time intravenous (IV) infusion or intrathecal (IT) injection. Dosage determined by participant weight.
  Other Names: Zolgensma

SUMMARY:
This is a global, prospective, multi-center study that is designed to assess the long-term safety and efficacy of OAV101 in patients who participated in an OAV101 clinical trial. The assessments of safety and efficacy in Study COAV101A12308 will continue for 5 years after enrollment in this study.

DETAILED DESCRIPTION:
The study is comprised of a Baseline Visit and 2 Follow-up Periods. For Follow-up Periods 1 and 2, which includes Baseline through Year 5 visits, assessments will be performed at the Investigational site. For the first 2 years (Follow-up Period 1), visits will occur every 6 months. For Years 3 to 5 (Follow-up Period 2) follow-up visits will be conducted annually. All patients will enter the study at the baseline visit and continue for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participated in an OAV101 clinical trial.
2. Written informed consent must be obtained before any assessment is performed.
3. Patient/Parent/legal guardian willing and able to comply with study procedures.

Exclusion Criteria:

There are no exclusion criteria for this study.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2030-09-26 (Estimated); Study Completion 2031-02-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent serious adverse events (SAEs) | Up to Year 5
  An SAE is defined as any adverse event [appearance of (or worsening of any pre-existing)] undesirable sign(s), symptom(s), or medical conditions(s) which meets any one of the following criteria:
  * fatal
  * life-threatening
  * results in persistent or significant disability/incapacity
  * constitutes a congenital anomaly/birth defect, fetal death or congenital abnormality or birth defect
  * requires in-patient hospitalization or prolongation of existing hospitalization, unless hospitalization is for routine treatment or monitoring of the studied indication, not associated with any deterioration in condition
  * is medically significant, e.g. defined as an event that jeopardizes the participant or may require medical or surgical intervention to prevent one of the outcomes listed above
Number of participants with treatment emergent Adverse Events of Special Interest (AESI) | Up to Year 5
  The following are important identified and important potential risks (AESI) associated with OAV101: Hepatotoxicity, Transient Thrombocytopenia, Cardiac adverse events, Sensory abnormalities suggestive of ganglionopathy, and Thrombotic microangiopathy. These will be assessed by the investigator.

SECONDARY OUTCOMES:
The number of participants demonstrating each developmental milestone according to the Developmental Milestone Checklist | Up to Year 5
  The Developmental Milestone Checklist is a sponsor created list of items using relevant definitions obtained from World Health Organization Multicentre Growth Reference Study (WHO-MGRS). These will be assessed via the milestone checklist, formed of 6 yes/no questions. The developmental milestones are: sitting with support, hands-and-knees crawling, standing with assistance, walking with assistance, standing alone and walking alone. A yes response indicates that the patient reached a particular development milestone.
The number of participants demonstrating maintenance of each developmental milestone according to the Developmental Milestone Checklist | Up to Year 5
  The Developmental Milestone Checklist is a sponsor created list of items using relevant definitions obtained from World Health Organization Multicentre Growth Reference Study (WHO-MGRS). These will be assessed via the milestone checklist, formed of 6 yes/no questions. The developmental milestones are: sitting with support, hands-and-knees crawling, standing with assistance, walking with assistance, standing alone and walking alone. A yes response indicates that the patient reached a particular development milestone.
Change from Baseline in the Hammersmith Functional Motor Scale - Expanded (HFMSE) total score | Up to Year 5
  The HFMSE is a validated SMA specific assessment devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.
Change from Baseline in the Revised Upper Limb Module (RULM) total score | Up to Year 5
  The RULM is a validated SMA specific assessment of motor performance in the upper limbs from childhood through adulthood in ambulatory and non-ambulatory individuals with SMA. The scale consists of 19 scorable items: 18 items scored on 0 (unable) to 2 (full achievement) scale, and one item that is scored from 0 (unable) to 1 (able). Total scores range from 0-37 points. Higher scores reflect higher level of motor ability.
Systolic and diastolic blood pressure (mmHg) | Up to Year 5
Number of patients with potentialy clinically significant vital sign findings - Respiratory Rate (breaths/min) | Up to Year 5
Number of patients with potentialy clinically significant vital sign findings -Pulse Rate (beats/min) | Up to Year 5
Number of patients with potentialy clinically significant vital sign findings -Temperature (Degrees Celsius) | Up to Year 5
Number of patients with potentialy clinically significant vital sign findings -Oxygen saturation level (%). | Up to Year 5
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated+saturated) in the blood and then multiplied by 100.

CONTACTS AND LOCATIONS:
Locations (29):
- Child Hosp Of The Kings Daughters, Norfolk, Virginia, United States
- Novartis Investigative Site, Sydney, New South Wales, Australia
- Novartis Investigative Site, Leuven, Belgium
- Brazil (2):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Montreal, Quebec, Canada
- China (4):
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Copenhagen, Denmark
- France (4):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Garches
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Roma, RM, Italy
- Japan (2):
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Spain
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/